CLINICAL TRIAL: NCT02890264
Title: Monitoring the Quality of Life of Patients With End-stage Renal Disease (QV-REIN) - Dialysis
Brief Title: Monitoring the Quality of Life of Patients With End-stage Renal Disease (QV-REIN)
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Quality of Life
Keywords: End stage renal disease; Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose for holding this survey is epidemiological surveillance, it must provide the indicators that contribute to the evaluation of the plan "improvement of the quality of life in chronic diseases" and monitoring the goal of 81 health law public in August 2004. This survey is intended to be renewed during the implementation period of the public health law to provide plan monitoring indicators.

The main objective is : To describe the quality of life of patients with major end-stage renal disease treated with dialysis method for at least one year.

The seconds objectives are :

* To contribute to the knowledge of the key determinants of the quality of life among chronic renal failure patients.
* To study the influence on way of giving a questionnaire about assessment of level of quality of life

DETAILED DESCRIPTION:
The proposed scheme is that of a repeated cross-sectional survey, with prevalent patients dialysis for at least 1 year, by self-administered questionnaires using standardized instruments and passed among a representative sample of subjects included in the nine participating regions kidney system. The first study in 2005, it is required to be repeated during the plan period (theoretically in 2007, 2009 and 2011).

Three studies will be carried out between 2005 and 2010. The progress of each study is the same.

The random draw of eligible patients, according to a stratification by region and age group is carried out by the Biostatistics and Medical Informatics Service of the Necker Hospital in Paris, responsible for basic SIMS-REIN, for data center in the regions Champagne-Ardenne, Languedoc-Roussillon, Limousin and Provence-Alpes-Côte d'Azur. For Auvergne, Bretagne, Lorraine and Rhône-Alpes, which operate independently for the collection of data REIN, the random draw of patients is done by each epidemiological center responsible for this collection.

The Biostatistics and Medical Informatics Service of the Necker Hospital, and epidemiological centers of Auvergne, Bretagne, Lorraine and Rhône Alpes must submit the list of selected patients Clinical Research Associate (CRA) national.

ELIGIBILITY:
Inclusion Criteria:

* Patient prevalent dialysis for at least 1 year
* Age at least 18 years old at the time of dialysis at
* Treaty within one of the nine aforementioned regions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The source population is all patients included in the REIN system at the time of the survey in the nine participating regions currently in the system: Auvergne, Bretagne, Centre, Champagne Ardennes, Languedoc Roussillon, Limousin, Lorraine, Provence Alpes Côte d 'Azur, Rhône Alpes.
  The patients selected to participate in the study were selected by random draw on all of the base, from those whose annual spot date falls during the investigation period.
  The random draw is stratified by region and age group with a sampling fraction proportional to the size of the original population.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
quality of life questionnaire for patients with end-stage renal disease | Every two years during six years

SECONDARY OUTCOMES:
mode of quality of life questionnaire administration | After one year of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Serge BRIANCON, Principal Investigator — Central Hospital Nancy

IPD SHARING:
Plan to Share IPD: No